CLINICAL TRIAL: NCT02276248
Title: Radiotherapy Combined With GDP (Gemcitabine, Cisplatin, Dexamethasone) Chemotherapy in Stage I/II Extranodal Natural Killer/T-cell Lymphoma Patients With Unfavorable Prognostic Factors: an Open-label, Single-arm, Phase II Clinical Trial
Brief Title: Radiotherapy Combined With GDP Chemotherapy in Stage I/II Extranodal Natural Killer/T-cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mei Dong, Department of Medical Oncology, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GREEN
Record Dates: First submitted 2014-10-23; First posted 2014-10-28 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Stage I/II Extranodal NK/T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- radiotherapy+chemotherapy (Experimental): Radiotherapy technique: Intensity-modulated radiation therapy total dose: 50 to 56 grays per fraction: 2 grays GDP chemotherapy: gemcitabine (1000mg/m2 intravenously over 30 minutes on days 1 and 8), cisplatin (25mg/m2 intravenously over 60 minutes on days 1-3), and dexamethasone (20mg/d orally on days 1-4 and days 11-14), which was administered every 21 days.
  Interventions: Radiation: Intensity-modulated radiation therapy; Drug: GDP chemotherapy

INTERVENTIONS:
Radiation: Intensity-modulated radiation therapy — total dose: 50 to 56 grays per fraction: 2 grays
Drug: GDP chemotherapy — gemcitabine (1000mg/m2 intravenously over 30 minutes on days 1 and 8), cisplatin (25mg/m2 intravenously over 60 minutes on days 1-3), and dexamethasone (20mg/d orally on days 1-4 and days 11-14), which was administered every 21 days.

SUMMARY:
This study is to evaluate the efficacy and safety of radiotherapy combined with GDP (gemcitabine, cisplatin, dexamethasone) chemotherapy in stage I/II extranodal natural killer/T-cell lymphoma patients with unfavorable prognostic factors.

DETAILED DESCRIPTION:
Radiotherapy has been recognized as the definitive treatment of choice for stages I and II extranodal NK/T cell lymphoma. The progression-free survival rate and overall survival rate of radiotherapy plus anthracycline-containing chemotherapy were comparable to that of radiotherapy alone. Our previous studies demonstrated the high responsiveness and safety of GDP (gemcitabine, cisplatin, dexamethasone) regimen in patients with extranodal NK/T cell lymphoma. Therefore, we design this study to evaluate the safety and benefit of radiotherapy plus GDP regimen in extranodal NK/T cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of ENKTL with typical morphology and immunophenotype according to the 2008 World Health Organization classification of lymphomas;
2. newly-diagnosed patients;
3. tumors primarily occurring in the upper aerodigestive tract (nasal cavity, nasopharynx, oral cavity, oropharynx and hypopharynx);
4. Ann Arbor stage I/II;
5. age ≥ 18 years;
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-2;
7. at least one measurable lesion;
8. adequate hematologic, hepatic, and renal functions: absolute neutrophil count ≥ 1.5×109/l, platelet count ≥ 100×109/l, total bilirubin ≤ 1.5 × upper limit of normal, AST and ALT ≤ 2 × upper limit of normal, and creatinine ≤ 1.5 mg/dl;
9. with at least one unfavorable prognostic factor (age > 60 years; B symptoms; elevated lactate dehydrogenase; regional node involvement; local tumor invasion: bone or skin; histologic elevation of high Ki-67 staining)
10. life expectancy of more 3 months;
11. informed consent.

Exclusion Criteria:

1. patients who received prior treatment;
2. stage I/II patients without unfavorable prognostic factors;
3. tumors primarily occurring in the extra-upper aerodigestive tract (e.g., skin, testis, intestine, muscle and so on);
4. pregnant or breastfeeding women and women of childbearing potential not employing adequate contraception;
5. patients with second primary cancer (except, adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumors curatively treated with no evidence of disease for ≥5 years)
6. patients with defect of central nervous system (CNS) or any psychiatric disorders and CNS metastases
7. other serious illness or medical conditions A. Clinically significant cardiac disease (uncontrolled congestive heart disease despite treatment [NYHA class III or IV], symptomatic coronary artery disease, unstable angina or myocardial infarction, conduction abnormality like grade 2 AV block, serious arrhythmia needed for medication, uncontrolled hypertension) within 6 months prior to study entry B. Liver cirrhosis (≥ Child-Pugh class B) C. History of significant neurologic or psychiatric disorders including dementia or seizures D. Active uncontrolled infection E. Other serious underlying medical conditions which could impair the ability of the patient to participate in the study
8. systemic anticancer therapy within 30 days before inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
2-year progression-free survival | 2 year

SECONDARY OUTCOMES:
2-year overall survival | 2 year
number of patients with adverse events | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Mei Dong, Principal Investigator — Cancer Hospital and Institute, Chinese Academy of Medical Sciences (CAMS) and Peking Union Medical College (PUMC)
Locations (1):
- Cancer Hospital and Institute, Chinese Academy of Medical Sciences (CAMS) and Peking Union Medical College (PUMC), Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Qi F, Wang WH, He XH, Chen B, Gui L, Fang H, Liu P, Wang SL, Yang JL, Song YW, Yang S, Qi SN, Zhou SY, Li YX, Dong M. Phase 2 Study of First-line Intensity Modulated Radiation Therapy Followed by Gemcitabine, Dexamethasone, and Cisplatin for High-Risk, Early Stage Extranodal Nasal-Type NK/T-Cell Lymphoma: The GREEN Study. Int J Radiat Oncol Biol Phys. 2018 Sep 1;102(1):61-70. doi: 10.1016/j.ijrobp.2018.05.046. Epub 2018 May 29. PMID 30102205